CLINICAL TRIAL: NCT01903629
Title: A Double-center Self-controlled Comparative Study of the Magnetic-controlled Capsule Endoscopy Versus Standard Gastroscopy for Gastric Diseases
Brief Title: Comparative Study of the Magnetic-controlled Capsule Endoscopy Versus Standard Gastroscopy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Second Military Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AKE-1
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Gastric Symptoms; Indicated for Upper GI Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- magnetic-controlled capsule endoscocpy (MCE) (Experimental): patients were assigned to swallow MCE first, followed by the gastroscopy
  Interventions: Device: MCE; Device: Standard gastroscopy

INTERVENTIONS:
Device: MCE — MCE first, followed by standard gastroscopy
Device: Standard gastroscopy

SUMMARY:
Passive video capsule endoscopy is the criterion standard for small-bowel diseases but cannot be used for the large gastric cavity.This blinded prospective study investigates the accuracy of the magnetic-controlled capsule endoscopy compared to gastroscopy in patients with gastric symptoms and indication for upper GI Endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric symptoms and indicated for Upper GI endoscopy
* Age of 18 years to 70 years

Exclusion Criteria:

* Patients with impaired bowel movement from ileus or organic digestive diseases
* Patients with known large and obstructing tumors of the upper GI tract
* Patients after upper GI surgery or abdominal surgery altering GI anatomy
* Patients under full anticoagulation
* Patient in poor general condition
* Patients using equipment that may be affected by radio transmission
* Patients using equipment that may be affected by magnetic field
* Pregnancy or suspected pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of magnetic-controlled capsule endoscopy(MCE) Versus Standard Gastroscopy in the diagnosis of diffuse and local lesions | 2 days

SECONDARY OUTCOMES:
Examination times of capsule and standard gastroscopy | 1 hour
Patient acceptance of capsule gastroscopy and standard gastroscopy | 3 days
Adverse events of both procedures | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

REFERENCES:
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Derived] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177